CLINICAL TRIAL: NCT00314717
Title: The Effect of a Low Glycemic Index Diet on Blood Sugar Control in Women With Gestational Hyperglycemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Protocol reference 16929
Record Dates: First submitted 2006-04-13; First posted 2006-04-14 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2007-08

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Control diet
Behavioral: Low GI diet

SUMMARY:
The purpose of the study is to see if a low glycemic index diet will reduce blood sugar levels in pregnant women with high blood sugar levels.

DETAILED DESCRIPTION:
Women with gestational hyperglycemia, including women with gestational diabetes and impaired glucose tolerance of pregnancy, consuming a low glycemic index (GI) diet will experience better blood glucose control thereby decreasing the risk associated complication(s).

ELIGIBILITY:
Inclusion Criteria:

* women with gestational hyperglycemia
* age between 18 and 45 inclusive
* willing and able to comply with protocol

Exclusion Criteria:

* <18 or >45 years of age
* other chronic or acute illness which affects carbohydrate metabolism
* known multiple pregnancy
* >34 weeks gestation
* language barrier (no translator available)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2006-04; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Fasting serum glucose | Baseline and 4 weeks
A1c | Baseline and 4 weeks
Self-blood-glucose-monitoring results | daily until delivery

SECONDARY OUTCOMES:
maternal weight gain throughout pregnancy | weekly
number of individuals who receive insulin treatment while participating in the study | duration of pregnancy
latency to insulin requirement/ gestational age when prescribed insulin | duration of pregnancy
dosage and frequency of insulin | duration of pregnancy
ultrasound measurements (if available) | according to clinical practice
fasting lipids | Baseline and 4 weeks
fasting c-reactive protein | Baseline and 4 weeks
infant birth weight | at birth
infant blood glucose | at birth
infant plasma calcium | at birth
infant bilirubin at birth obtained via heel prick | at birth
birth complications | at birth
perceptions of educational materials
perceptions of diet treatments

CONTACTS AND LOCATIONS:
Overall Officials: Thomas MS Wolever, MD, PhD, Principal Investigator — University of Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Grant SM, Wolever TM, O'Connor DL, Nisenbaum R, Josse RG. Effect of a low glycaemic index diet on blood glucose in women with gestational hyperglycaemia. Diabetes Res Clin Pract. 2011 Jan;91(1):15-22. doi: 10.1016/j.diabres.2010.09.002. Epub 2010 Nov 20. PMID 21094553